CLINICAL TRIAL: NCT02325440
Title: A 32-week, Monocentric, Exploratory, Single Arm Study to Assess Immune Function and MRI Disease Activity in Patients With RRMS Transferred From Previous Treatment With Natalizumab to Gilenya® (Fingolimod)
Brief Title: Study to Assess Immune Function and MRI Disease Activity in RRMS Patients When Switching From Natalizumab to Gilenya
Acronym: ToFingo2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM12_0037; 2013-004616-21 (EudraCT Number); CFTY720D2415T (Other: Novartis)
Record Dates: First submitted 2014-09-04; First posted 2014-12-25 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: RRMS (relapsing remitting multiple sclerosis); Cluster of differentiation 49d (CD49d); immune function; disease activity
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride; Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natalizumab - Washout - Fingolimod (Experimental): One experimental arm: Patients receive one final dose of natalizumab 300mg followed by an 8-week washout Phase and subsequent 32-week treatment Phase with fingolimod 0.5mg o.i.d.
  Interventions: Drug: Fingolimod; Drug: Natalizumab

INTERVENTIONS:
Drug: Fingolimod — Fingolimod: 0.5 mg p.o. (o.i.d)
  Other Names: FTY720; Gilenya
Drug: Natalizumab — Natalizumab: 300 mg i.v. (once at baseline);
  Other Names: Tysabri

SUMMARY:
A trial in patients with relapsing remitting multiple sclerosis (RRMS)

Main objectives:

* To evaluate changes in the reconstitution of immune surveillance over time upon switching from natalizumab to fingolimod assessed by a change in the expression of CD49d.
* To evaluate changes in the migratory capacity of immune cells/peripheral blood mononuclear cells (PBMCs) upon switching from natalizumab to fingolimod in an in-vitro model of the blood-brain-barrier (BBB).
* To evaluate changes in paraclinical disease activity over time upon switching from natalizumab to fingolimod assessed by MRI (changes in Gd+, T2w lesions and DTI).
* To evaluate changes in T1w / FLAIR lesions upon switching from natalizumab to fingolimod.

DETAILED DESCRIPTION:
Patients are screened and must sign informed consent at visit 1. At the 2nd visit, all patients receive a baseline infusion of Natalizumab, which is followed by an 8 week washout Phase. After the washout Phase all patients receive fingolimod for 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male and female subjects aged 18-65 yrs.
3. Subjects with RRMS, defined by 2010 rev. McDonald criteria.
4. Patients with an (EDSS) score of 0-6.0 inclusive.
5. Patients on treatment with natalizumab for ≥ 12 months prior to screening where treatment discontinuation is considered for any of the following reasons:

   * treatment duration for more than 2 years
   * positive JC virus (JCV) antibody status
   * adverse effects including hypersensitivity reactions
   * presence of anti-natalizumab neutralizing antibodies
   * any other valid medical reason

Exclusion Criteria:

1. Patients with a history of chronic disease of the immune system other than MS, which requires systemic immunosuppressive treatment, or a known immunodeficiency syndrome.
2. Patients with Crohn´s disease or ulcerative colitis.
3. Patients who have been treated with:

   * systemic corticosteroids or immunoglobulins within 1 month prior to baseline.
   * immunosuppressive medications such as azathioprine, cyclophosphamide or methotrexate within 3 months prior to baseline.
   * monoclonal antibodies (excluding natalizumab) within 3 months prior to baseline.
   * cladribine or mitoxantrone at any time.
4. History of malignancy of any organ system (other than cutaneous basal cell carcinoma).
5. Uncontrolled diabetes mellitus (HbA1c >7%).
6. Diagnosis of macular edema during Screening Phase.
7. Severe active infections, active chronic infection.
8. Negative for varicella-zoster virus immunoglobulin G antibodies prior to baseline.
9. Patients that received any live or live-attenuated vaccine (including varicella-zoster virus or measles) within 1 month prior to baseline.
10. Patients who have received total lymphoid irradiation or bone marrow transplantation.
11. Patients with any medically unstable condition, as assessed by the investigator.
12. Patients with certain cardiovascular conditions and/or findings in the screening ECG.
13. Patients with certain lung diseases.
14. Patients with certain hepatic conditions.
15. Patients with a screening white blood cell (WBC) count <3,500/mm3 or lymphocyte count <800/mm3.
16. Patients with certain neurologic/psychiatric disorders:
17. Patients unable to undergo MRI scans, including claustrophobia or history of hypersensitivity to gadolinium-diethylenetriaminepentacetate (Gd-DTPA).
18. Patients who have received an investigational drug or therapy within 180 days or 5 half-lives before baseline, whichever is longer.
19. Pregnant or nursing (lactating) women, confirmed by a positive human chorionic gonadotropin laboratory.
20. Women of child-bearing potential unless they are using effective contraception during the study and for 5 half-lives after stopping treatment. In case of use of oral contraception women should have been stable on the same medication for a minimum of 3 months before baseline.
21. History of hypersensitivity to the study drugs or to drugs of similar chemical classes.
22. Prior participation in a trial with fingolimod.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Temporal changes in the expression of CD49d | weeks: 12, 16, 20, 24, 28, 32
  First Co-Primary Objective; Flow-cytometric analysis of temporal changes in the expression of CD49d of PBMCs; unit of measure: mean fluorescence intensity (MFI)
Migratory capacity of immune cells | weeks: 12, 32
  Second Co-Primary Objective; in-vitro model of the blood-brain-barrier (BBB) with subsequent flow-cytometric analysis and bead based quantification assessing temporal changes in the migratory capacity of immune cells; unit of measure: fluorescence intensity

SECONDARY OUTCOMES:
MRI disease activity over time by GD+, T2w and DTI | weeks: 0, 8, 12, 16, 24, 32
  Number of active (new or newly enlarging) lesions are assessed over time by MRI (changes in Gadolinium (GD+), T2w lesions and DTI (Diffusion Tensor Imaging))
MRI disease activity over time by T1w / FLAIR | weeks: 0, 8, 12, 16, 24, 32
  Number of active (new or newly enlarging) lesions are assessed over time by MRI (T1w / FLAIR (Fluid Attenuated Inversion Recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Klotz, PD. Dr. med., Principal Investigator — Universitätsklinikum Muenster, Germany
Locations (1):
- Universitaetsklinikum Muenster, Department of Neurology, Münster, Germany

REFERENCES:
- [Derived] Lohmann L, Janoschka C, Schulte-Mecklenbeck A, Klinsing S, Kirstein L, Hanning U, Wirth T, Schneider-Hohendorf T, Schwab N, Gross CC, Eveslage M, Meuth SG, Wiendl H, Klotz L. Immune Cell Profiling During Switching from Natalizumab to Fingolimod Reveals Differential Effects on Systemic Immune-Regulatory Networks and on Trafficking of Non-T Cell Populations into the Cerebrospinal Fluid-Results from the ToFingo Successor Study. Front Immunol. 2018 Jul 9;9:1560. doi: 10.3389/fimmu.2018.01560. eCollection 2018. PMID 30050529